CLINICAL TRIAL: NCT04580784
Title: Weekly Single Fraction Hypofractionated Adjuvant Radiotherapy for Early Stage Breast Cancer: A Single Institution Feasibility Study
Brief Title: Weekly Single Fraction Hypofractionated Adjuvant Radiotherapy for Early Stage Breast Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mona Salem (Other)
Collaborators: Kasr El Aini Hospital (Other)
Responsible Party: Sponsor-Investigator, Mona Salem, Assistant Lecturer of clinical oncology, Kasr El Aini Hospital
Organization: Kasr El Aini Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FAST feasibility in CU
Record Dates: First submitted 2019-06-07; First posted 2020-10-08 (Actual); Last update posted 2020-10-08 (Actual); Status verified 2020-10

CONDITIONS: Breast Cancer; Radiotherapy Side Effect
Keywords: Breast cancer; Radiotherapy; Hypofractionation
MeSH Terms: conditions — Breast Neoplasms; Radiation Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Hypofractionation (Experimental): Hypofractionated whole breast radiotherapy using a dose of 28.5 Gy over 5 fractions with once weekly fractions.
  Interventions: Radiation: Weekly hypofractionation for early breast cancer

INTERVENTIONS:
Radiation: Weekly hypofractionation for early breast cancer — Testing the feasibility of a hypofractionated adjuvant radiotherapy regimen after breast surgery on a-once-weekly basis for a total dose of 28.5Gy in 5 fractions over 5 weeks

SUMMARY:
The current study is a prospective phase II study; Eligible patients will receive hypofractionated Irradiation at a total dose of 28.5Gy in 5 once-weekly fractions of 5.7Gy in 5 weeks to the Whole Breast or chest wall with or without peripheral lymphatic irradiation.

DETAILED DESCRIPTION:
Testing the feasibility of a hypofractionated adjuvant radiotherapy regimen after breast surgery on a-once-weekly basis for a total dose of 28.5Gy in 5 fractions over 5 weeks in Kasr EL Aini Hospital.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically proven diagnosis of invasive breast adenocarcinoma.
2. Prior radical surgery (Modified Radical Mastectomy or Breast Conservative Surgery).
3. No macroscopic evidence of distant metastases at diagnosis.

Exclusion Criteria:

1. Prior radiation to the thoracic region.
2. Pregnancy.
3. Patients with synchronous or prior malignancy.
4. Positive surgical margins.

Min Age: 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 20 (Estimated)
Dates: Start 2018-12-10 (Actual); Primary Completion 2020-11 (Estimated); Study Completion 2024-05 (Estimated)

PRIMARY OUTCOMES:
Change in cosmetic breast appearance | six months
  according to HARVARD cosmesis scale: 1 Excellent, 2Good, 3 Fair and 4 Poor
Acute radiation toxicity assessment | six months
  according to the RTOG acute toxicity scale: 0 No visible change, 1 faint/dull erythema, 2tender/ bright +- dry desquamation, 3 patchy moist desquamation, 4 conflueunt moist desquamation, pitting edema, 0 is the best and 4 is the worse.
Patient quality of life assessment. | six months
  according to FACT-B
Patient satisfaction. | six months
  according to FACIT-TS-PS

CONTACTS AND LOCATIONS:
Overall Officials: Mona Salem, MSc, Principal Investigator — Kasr El AiniH
Locations (1):
- Kasr El AiniH, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No